CLINICAL TRIAL: NCT05463913
Title: Ultra-long Field-Of-View Positron Emission Tomography for Characterization of Indeterminate Lung Nodules: a Pilot Study Exploring Opportunities for Clinical Research
Brief Title: Lung Nodule Detection Using Ultra-long FOV PET/CT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 202100174
Record Dates: First submitted 2022-03-22; First posted 2022-07-19 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Blinded for FDG PET/CT conducted for research results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 18F-FDG — Patients will receive a single intravenous injection of 3 MBq/kg 18F-FDG
Radiation: PET/CT imaging — Patient will undergo 2 CT acquisitions and multiple PET emission scans.

SUMMARY:
Indeterminate lung nodules (6-15mm) are frequent findings in patients undergoing chest CT scanning, but adequate follow-up imaging is currently not in place to facilitate early detection, diagnosis and decision making regarding treatment.

The introduction of long Field-Of-View PET/CT scanners could make a difference in this matter due to the substantial increase in sensitivity allowing optimal image quality. Whether this new technology could provide improved detection and follow-up of indeterminate lung nodules is what we aim to explore in this study.

DETAILED DESCRIPTION:
Indeterminate lung nodules (6-15 mm) are frequent findings in patients undergoing chest Computed Tomography (CT). In the large randomized controlled Dutch-Belgian lung cancer screening trial NELSON, overall, 9.2% of the screened participants had an initially indeterminate CT scan. To decrease mortality from lung cancer, early identification of malignant lesions among the many lung nodules is crucial. The probability of malignancy depends on size and other factors. It is difficult to determine whether a nodule is malignant on size alone. For further differentiation of a lung nodule, usually, repeated chest CT scanning is performed at 3-6 months up to 2 years to assess nodule growth, and/or 2-deoxy-2-[fluorine-18) fluoro-D-glucose (18F-FDG) Positron Emission Tomography (PET)/CT to evaluate metabolic activity. However, repetitive CT scans are not favoured because of radiation exposure, patiënt anxiety, and potential delay in cancer diagnosis. Furthermore, 18F-FDG PET/CT has thus far insufficiënt sensitivity for detection and characterization of small (in particular < 1 cm) lung nodules, meaning that a negative result does not rule out the presence of cancer, which thus usually requires further follow-up CT scans. Improvement in work-up of indeterminate lung nodules is urgently needed, in particular with the expected introduction of lung cancer screening in the coming years.

In this study, the aim is to derive optimal imaging procedures and to assess the technical performance of the Vision Quadra PET/CT system concerning its feasibility to detect indeterminate lung nodules. Furthermore, this study aims to preliminary explore the sensitivity, specificity, and accuracy of the characterisation of lung nodules using the Vision Quadra PET/CT.

After enrolment, patients will receive a Standard 3 MBq/kg injection of 18F-FDG and undergo whole-body dynamic PET/CT acquisition at 30-60 min post-injection (pi), followed by a 10 min whole-body list-mode PET/CT acquisition. Subsequently, patients will be asked to hold their breath for 15 seconds to assess the added value of a single fast deep-inspiration breath-hold acquisition.

At 120 min pi a second 10 min whole-body list-mode PET/CT will be acquired to potentially further differentiate between inflammation and malignancy.

The list-mode acquisitions can be reprocessed retrospectively with less counts to produce images representing scans collected with lower activity administration or shorter scan times (e.g., a 1 min instead of 10 min PET scan is equivalent to 10% of the injected activity at scan start). Quantitative image analysis results will be correlated with pathology (benign or malignant) of the lung lesion, and results of a previously performed routine-care 18F-FDG PET/CT and CT chest.

ELIGIBILITY:
Inclusion Criteria:

* able to give informed consent
* signed informed consent
* confirmed indeterminate lung nodule(s) of 6-15 mm in size on CT chest imaging
* routine 18F-FDG PET/CT performed
* scheduled for biopsy or resection of the lung nodules

Exclusion Criteria:

* claustrophobia
* pregnant or breastfeeding
* interval of at least 2 weeks between PET scan and last date of systemic anti-cancer therapy to reduce false-negative uptake in lesions
* radiation therapy of the target lung nodule(s)
* uncontrolled diabetes mellitus
* any medical condition potentially hampering conduction of the trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Description of optimized (in terms of e.g. activity dose needed for injection, time of scan duration, post-processing filtering) static whole-body acquisition and reconstruction protocol by performing semi-quantitative (SUV) analysis. | up to 2 years
  Description of optimized (in terms of e.g. activity dose needed for injection, time of scan duration, post-processing filtering) static whole-body acquisition and reconstruction protocol by performing semi-quantitative (SUV) analysis.
Description of optimized (in terms of e.g. activity dose needed for injection, time of scan duration) dynamic whole-body acquisition and reconstruction protocol by performing kinetic modelling (Patlak, Ki) analysis. | up to 2 years
  Description of optimized (in terms of e.g. activity dose needed for injection, time of scan duration) dynamic whole-body acquisition and reconstruction protocol by performing kinetic modelling (Patlak, Ki) analysis.
Description of optimized breath-hold acquisition and reconstruction protocol by performing semi-quantitative (SUV) analysis and compare with outcomes 1 and 2. | up to 2 years
  Description of optimized breath-hold acquisition and reconstruction protocol by performing semi-quantitative (SUV) analysis and compare with outcomes 1 and 2.

SECONDARY OUTCOMES:
Inventory of early detection and possibly characterization of indeterminate lung nodules | up to 2 years
  (i.e., to distinguish between benign and malignant tissue) including preliminary exploration of sensitivity, specificity, and accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne H Brouwers, MD PhD, Principal Investigator — Nuclear Medicine physician
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No